CLINICAL TRIAL: NCT06450275
Title: Randomized, Two-way, Two-period, Single Oral Dose, Open-label, Crossover, Bioequivalence Study to Compare Dolutegravir 50mg Film-coated Tablets (50mg Dolutegravir) Versus Tivicay 50mg Film-coated Tablets (50mg Dolutegravir) in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study to Compare Dolutegravir 50mg Film-coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1233-2023
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dolutegravir Film Coated Tablet (Experimental): Dolutegravir 50mg Film Coated Tablet
  Interventions: Drug: Dolutegravir 50 MG Film Coated Tablet
- Tivicay film-coated tablets (Active Comparator): Tivicay 50mg, film-coated tablets
  Interventions: Drug: Tivicay 50mg, film-coated tablets

INTERVENTIONS:
Drug: Dolutegravir 50 MG Film Coated Tablet — 1 tablet of Dolutegravir 50mg film-coated tablets
  Arms: Dolutegravir Film Coated Tablet
Drug: Tivicay 50mg, film-coated tablets — 1 tablet of Dolutegravir 50mg film-coated tablets
  Arms: Tivicay film-coated tablets

SUMMARY:
Randomized, two-way, two-period, single oral dose, open-label, crossover, bioequivalence study to compare Dolutegravir 50mg film-coated tablets (50mg Dolutegravir) versus Tivicay 50mg film-coated tablets (50mg Dolutegravir) in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

A. The subject is Caucasian & aged between eighteen & fifty years (18 - 50), both inclusive.

B. The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 30.0kg/m2). C. The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.

D. The results of medical history, physical examination, vital signs & conducted medical laboratory tests are normal as determined by the clinical investigator. E. The subject tested negative for Hepatitis B (HBsAg), Hepatitis C (HCVAb) and human immunodeficiency virus (HIVAb). F. There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements. G. The subject is able to understand and willing to sign the informed consent form.

H. For female subjects: negative serum pregnancy test and the woman is using two reliable contraception methods and not lactating. I. The subject has normal cardiovascular system & normal ECG with normal QT interval corrected for heart rate according to Bazett's formula. J. The subject's kidney and liver (AST & ALT enzymes) function tests are within normal range.

(Creatinine is accepted if below the reference range after being evaluated by the CI as clinically not significant).

Exclusion Criteria:

A. The subject is a heavy smoker (more than 10 cigarettes per day). B. The subject has suffered an acute illness one week before dosing. C. The subject has a history of or concurrent abuse of alcohol. D. The subject has a history of or concurrent abuse of illicit drugs. E. The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.

F. The subject has been hospitalized within three months before the study or during the study.

G. The subject is on special diet (for example subject is vegetarian). H. The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 72 hours after dosing in all study periods.

I. The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.

J. The subject has taken grapefruit/ orange containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.

K. The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.

L. The subject has donated blood within 80 days before first dosing. M. The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.

N. The subject has consumed drugs, herbal products or supplements that may affect pharmacological or pharmacokinetic properties of Dolutegravir (for example: Etravirine, Lopinavir, Ritonavir, Darunavir, Efavirenz, Nevirapine, Rilpivirine, Tenofovir, Atazanavir, Tipranavir, Fosamprenavir, Daclatasvir, Fampridine, Carbamazepine, Oxcarbazepine, Phenytoin, Phenobarbital, Ketoconazole, Fluconazole, Itraconazole, Posaconazole, Voriconazole, St.

John's wort, Magnesium/ Aluminium- containing antacid, Calcium supplements, Iron supplements, Multivitamin, Prednisone, Metformin, Rifampicin, Rifabutin, Ethinyl Estradiol, Norelgestromin, Zink & Methadone) two weeks before dosing, during the study and two weeks after dosing.

Note: Subjects, who were screened for another study and were not enrolled, might be recruited for this study provided they meet the acceptance criteria of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Maximum concentration obtained (Cmax) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data Cmax
AUC from time 0 to last collection time t (AUC0-t) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data AUC0-t

SECONDARY OUTCOMES:
AUC from time 0 to infinity (AUC0-inf) | 23 hours
  Description Statistics
  Description Statistics Description Statistics
Time of the maximum measured plasma concentration (Tmax) | 23 hours
  Description Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- ACDIMA Biocenter, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No